CLINICAL TRIAL: NCT04970563
Title: Detection of Asymptomatic SARS-Cov2 Infected Patients by Detection Dogs: "Proof of Concept" Study
Brief Title: Detection of Asymptomatic SARS-Cov2 Infected Patients by Detection Dogs: "Proof of Concept" Study (CoviDetectionDog)-Covid-19
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hôpital Européen Marseille (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 21-12
Record Dates: First submitted 2021-06-16; First posted 2021-07-21 (Actual); Last update posted 2022-04-14 (Actual); Status verified 2021-06

CONDITIONS: Infection by SARS-COV-2; Healthy Controls

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Patients infected by SARS-COV-2 (RT-PCR +) and asymptomatic (Experimental)
  Interventions: Other: Body odor samples
- "Control" group: patients infected by SARS-COV-2 (RT-PCR +) and symptomatic (Other)
  Interventions: Other: Body odor samples
- "Healthy controls" group: not infected by SARS-COV-2 (RT-PCR-) and asymptomatic. (Other)
  Interventions: Other: Body odor samples

INTERVENTIONS:
Other: Body odor samples — Participants will provide six body odor samples (mask and sweat samples) at inclusion
  Arms: "Control" group: patients infected by SARS-COV-2 (RT-PCR +) and symptomatic; Patients infected by SARS-COV-2 (RT-PCR +) and asymptomatic
Other: Body odor samples — Participants will provide six body odor samples (masks and compresses) at inclusion. A 7-day follow-up will be carried out to check, respectively, the absence of symptoms and the persistence of negativity on the SARS-COV-2 PCR test
  Arms: "Healthy controls" group: not infected by SARS-COV-2 (RT-PCR-) and asymptomatic.

SUMMARY:
The spread of the new SARS-CoV-2 virus has led to a pandemic. Described for the first time in China at the end of 2019, it causes Covid-19 disease. Its characteristics in terms of contagiousness and lethality have led countries to adapt their screening and care strategies.

Early and accurate identification of people infected with SARs-CoV-2 is an essential measure to confront Covid-19 pandemic. A key aspect of Covid-19 is that diagnostic tests must be able to detect the virus in asymptomatic, pre-symptomatic and symptomatic patients.

Changes in human odor, as symptoms of specific diseases, have been observed. Dogs have already been used to detect breast or lung cancer, diabetes, epilepsy or kidney disease with some success There is currently a growing body of research and previous work, though preliminary, indicating the possibility that dogs identify persons infected with Sars-Cov-2 compared to healthy persons.

The purpose of this study is to determine whether trained detection dogs are able to identify asymptomatic patients infected by Sars-Cov-2.

The investigators aim to validate the possibility to identify / discriminate patients with Covid-19 according to their odor by a proof of concept (with specificity and sensitivity of the detection test), i.e. new non-invasive screening method using dogs odor detection capabilities.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥ 18 years
* Having given free and informed written consent
* Being affiliated to the center national security system social
* Patients infected by SARS-COV-2 with positive RT PCR on nasopharyngeal swab and without symptoms (fever, cough, anosmia, diarrhea) will be included in "experimental" Group 1.
* Patients infected by SARS COV 2 with positive RT PCR on nasopharyngeal swab and presenting at least one symptom will be included in Group 2 "control".
* Participants not infected by SARS-COV-2 with negative RT PCR on nasopharyngeal sample and showing no symptoms on Day 0 and Day 7 will be included in Group 3 "healthy controls".

Exclusion Criteria:

- Patient whose life expectancy is less than 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2021-06-21 (Actual); Primary Completion 2022-01-14 (Actual); Study Completion 2022-01-14 (Actual)

PRIMARY OUTCOMES:
Percentage behavioral response of trained dogs obtained on sweat samples from patients infected by asymptomatic SARS-Cov-2. | Six months

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Européen Marseille, Marseille, France

IPD SHARING:
Plan to Share IPD: No